CLINICAL TRIAL: NCT00070967
Title: Effects of Acupuncture on Pain, Nausea, Quality of Life
Brief Title: Acupuncture to Improve Quality of Life in Patients With Advanced Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21AT001010-01 (NIH)
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Ovarian Cancer
Keywords: Acupuncture; Quality of Life; Complementary Therapies; TCM; Traditional Chinese Medicine
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
This study will test the feasibility of acupuncture as a complementary therapy for advanced cancer by comparing symptoms and quality of life before and after 8 weeks of acupuncture treatments.

DETAILED DESCRIPTION:
A large percentage of the practice and use of complementary and alternative medicine (CAM) in the United States is focused on cancer. Whether the CAM use is aimed at reducing one's risk of developing cancer or improving the quality of life of a cancer patient during treatment or at the end of life, the public focus on CAM and cancer has created a driving force for cancer centers to address the efficacy and science of these methods.

Currently, the majority of cancer patients do not receive adequate palliative care. Acupuncture has been shown to be effective in the treatment of pain and nausea and has also been shown to improve one's general well-being. Acupuncture also has some effectiveness in relieving symptoms of anxiety and depression. This study will evaluate the efficacy of acupuncture by Traditional Chinese Medicine clinicians to address the quality of life and symptoms of patients with incurable cancer.

Women with recurrent metastatic ovarian cancer and similar patients with advanced cancer who are ambulatory and receiving conventional palliative care will be enrolled in this study. Patients will continue to receive high-quality, conventional clinical interventions, including chemotherapy and pain and symptom reduction programs. Patients will also receive 8 weeks of acupuncture. Evaluation tools such as Satisfaction with Life Domains Scale for Cancer (SLDS-C), Brief Pain Inventory, and Rotterdam Symptom Check List will be used to assess the acupuncture intervention.

ELIGIBILITY:
Inclusion Criteria

* Advanced cancer patients, primarily ovarian cancer patients
* Undergoing palliative care treatment
* Ambulatory
* Symptomatic with pain, nausea, and/or an inadequate quality of life
* Platelets > 25,000/mm3
* ANC > 500 cells/mm3

Exclusion Criteria

* Acupuncture treatment during the 6 months prior to study entry
* History of bleeding disorder, such as hemophilia or von Willebrand disease
* Acute psychosis

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-09; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: David S. Rosenthal, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States